CLINICAL TRIAL: NCT00752700
Title: Resistance Training in Radically Treated Respiratory Cancer Patients: a Prospective Randomized Multicenter Study
Brief Title: Resistance Exercise Training For Radically Treated Respiratory Cancer
Acronym: REINFORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008/384
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Cancer
Keywords: Patients; radically; treated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Control group
- 2 (Active Comparator): Conventional resistance training program (CRT)
  Interventions: Other: Conventional resistance training
- 3 (Experimental): Whole body vibration resistance training (WBV) on the FITVIBE-platform
  Interventions: Other: Whole body vibration resistance training

INTERVENTIONS:
Other: Conventional resistance training — Conventional resistance training program (CRT)
  Arms: 2
Other: Whole body vibration resistance training — Whole body vibration resistance training (WBV) on the FITVIBE-platform
  Arms: 3

SUMMARY:
The first part of the study is an observational part. In eligible patients with early stage respiratory cancer, the primary and secondary endpoints will be evaluated before and after their scheduled radical cancer therapy. The measured variables, include a blood sample, pulmonary function tests, level of dyspnea, exercise tests, measurement of body composition, respiratory and peripheral muscle force, health related quality of life and psychological status. Only registered participants having completed a radical treatment and having either less than 70% of the predicted normal value of the quadriceps force (QF) or a decrease of more than 10% predicted value of the QF between pre-and post radical treatment, will be allowed to participate to the second part of the study. These patients will then be randomized in three groups. Group A, the control group, will have the usual care and follow up according to clinical symptoms. Group B will be offered a conventional resistance training program (CRT), and group C, will be offered a whole body vibration resistance training (WBV) on the FITVIBE-platform. All previous variables will be measured after 6 and 12 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-small cell or small cell lung cancer or mesothelioma candidate for radical treatment

  * either by surgical resection with or without perioperative chemotherapy
  * or by thoracic radiotherapy with or without chemotherapy
* Between 18 and 80 years of age
* Written informed consent

Supplementary criteria for PART II:

* Treatment for their cancer considered radical

  * either by surgical resection with or without perioperative chemotherapy
  * or by thoracic radiotherapy with or without chemotherapy
* having less than 70% of the predicted normal value of the Quadriceps Force (QF) or a decrease of more than 10% predicted value of the QF between the baseline and post-radical therapy measurement of QF
* Post treatment assessment maximum 14 days after radical treatment or between 6th and 8th week after radical treatment if the latter consists only of surgical resection

Exclusion Criteria:

Patients presenting with one or more of the following will be excluded:

* Severe anemia (Hb below 8 g/dl)
* Fever (> 38°C)
* Cachexia (loss of more than 35% of premorbid weight)
* Severe cardiac, neurological and orthopedic co-morbidity interfering with exercise training.
* A pacemaker, hip, knee of shoulder prosthesis or recently introduced spirals, metal pens, bolts or plates
* Uncontrolled diabetes, epilepsy or migraine
* Uncontrolled vertebral diseases (osteoporotic or metastatic fractures, acute hernia, discopathy, spondylitis)
* Open wounds

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The change of 6MWD observed between pre-and post radical treatment | 12 weeks
between post radical treatment and after a 12 week resistance training | 12 weeks

SECONDARY OUTCOMES:
The changes of the following variables: Muscle strength | 12 weeks
Muscle mass | 12 weeks
Body composition | 12 weeks
Maximal exercise capacity | 12 weeks
Muscle force | 12 weeks
Quality of life | 12 weeks
Anxiety and depression scores | 12 weeks
Dyspnea scores | 12 weeks
6MWD | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Meerbeeck, MD, PhD, Principal Investigator — University Hospital, Ghent; Eric Derom, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - AZ St. Jan, Bruges
  - CHU Saint Pierre, Brussels
  - University Hospital Ghent, Ghent
  - CHU Sart Tilman, Liège

REFERENCES:
- [Derived] Salhi B, Huysse W, Van Maele G, Surmont VF, Derom E, van Meerbeeck JP. The effect of radical treatment and rehabilitation on muscle mass and strength: a randomized trial in stages I-III lung cancer patients. Lung Cancer. 2014 Apr;84(1):56-61. doi: 10.1016/j.lungcan.2014.01.011. Epub 2014 Jan 23. PMID 24560331
- See also: Website of the University Hospital Ghent — http://www.uzgent.be